CLINICAL TRIAL: NCT01656395
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel-Group, Adaptive-Design, Dose-Ranging Study of MK-1029 in Adult Subjects With Persistent Asthma
Brief Title: A Dose-Ranging Study of MK-1029 in Adults With Persistent Asthma (MK-1029-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1029-012; 2012-000643-27 (EudraCT Number); 132230 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-07-03; First posted 2012-08-03 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- MK-1029 10 mg (Experimental): Participants receive MK-1029 10 mg tablets once daily (QD) for 12 weeks
  Interventions: Drug: MK-1029
- MK-1029 30 mg (Experimental): Participants receive MK-1029 30 mg tablets QD for 12 weeks
  Interventions: Drug: MK-1029
- MK-1029 60 mg (Experimental): Participants will receive MK-1029 two 30 mg tablets QD for 12 weeks
  Interventions: Drug: MK-1029
- MK-1029 150 mg (Experimental): Participants will receive MK-1029 150 mg tablets QD for 12 weeks
  Interventions: Drug: MK-1029
- Montelukast 10 mg (Active Comparator): Participants will receive Montelukast 10 mg tablets QD for 12 weeks
  Interventions: Drug: Montelukast 10 mg
- Placebo (Placebo Comparator): Participants will receive Placebo tablets QD for 12 weeks
  Interventions: Drug: Placebo
- MK-1029 1 mg or 3 mg (Experimental): Participants will receive either MK-1029 1 mg or 3 mg tablets (dose to be determined based on results of interim analysis from Part I) QD.
  Interventions: Drug: MK-1029
- Montelukast 10 mg + MK-1029 (Experimental): Participants will receive Montelukast 10 mg tablets QD and MK-1029 tablets (dose to be determined based on results of interim analysis from Part I) QD
  Interventions: Drug: Montelukast 10 mg

INTERVENTIONS:
Drug: MK-1029 — MK-1029 10 mg, 30 mg or 150 mg oral tablets taken QD at bedtime, based on randomization.
  Arms: MK-1029 1 mg or 3 mg; MK-1029 10 mg; MK-1029 150 mg; MK-1029 30 mg; MK-1029 60 mg
Drug: Montelukast 10 mg — Parts I-II: Participants will receive Montelukast 10 mg tablets QD
  Other Names: SINGULAIR®
  Arms: Montelukast 10 mg; Montelukast 10 mg + MK-1029
Drug: Placebo — Parts I-II: Participants will receive Placebo tablets QD
  Arms: Placebo

SUMMARY:
This adaptive design, dose-ranging study of MK-1029 will assess the dose-related efficacy and safety of MK-1029 compared with placebo using measures of lung function (forced expiratory volume in 1 second [FEV1]). The primary objectives are (1) To demonstrate that MK-1029, compared with placebo, results in dose-related improvements in FEV1 over the last 6 weeks of the 12-week active-treatment period; and (2) To determine the dose-related safety and tolerability of MK-1029 as monotherapy and as concomitant dosing with montelukast over 12 weeks. The primary hypothesis is: MK-1029 is superior to placebo in a dose-related fashion in the average change from baseline in FEV1 over the last 6 weeks of the 12-week active-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant or breastfeeding, and not planning to become pregnant during the study
* history of symptoms of persistent asthma for at least one year
* current use of acceptable asthma treatments and willingness to taper or discontinue these treatments; acceptable asthma treatments:

  * use of inhaled SABAs (e.g., albuterol/salbutamol) only "as-needed" with no use of asthma controller medications; OR
  * use of stable doses of low- or medium-dose inhaled corticosteroids (ICS), alone, or in combination with either a long-acting beta-agonist (LABA) or other asthma controller medications (including leukotriene receptor antagonists) and can tolerate tapering or discontinuation
* no history of smoking OR no smoking within <1 year with a smoking history of ≤10 pack-years
* ability to maintain a constant day/night, awake/sleep cycle
* agreement to not change habitual consumption of beverages or food containing caffeine throughout the study
* Body Mass Index (BMI) of 15 to 40 kg/m^2

Exclusion Criteria:

* myocardial infarction, congestive heart failure, or uncontrolled cardiac arrhythmia within past ≤3 months
* hospitalization within past ≤4 weeks
* major surgical procedure within past ≤4 weeks
* participation in a clinical study involving an investigational drug within past ≤4 weeks
* current regular use or recent (within past ≤5 years) past abuse of alcohol (>14 drinks/week) or illicit drugs
* donation of a unit of blood within past ≤2 weeks or intention to donate a unit of blood during the study
* evidence of another clinically significant, active pulmonary disorder such as chronic obstructive pulmonary disease (COPD)
* emergency room treatment for asthma within past ≤4 weeks or hospitalization for asthma within past ≤8 weeks
* respiratory tract infection requiring antibiotic treatment within past ≤8 weeks
* evidence of active, clinically significant sinus disease within past ≤1 week
* history of a clinically significant psychiatric disorder, other than stable depression, within past ≤12 weeks
* history of HIV
* hypersensitivity or intolerance to inhaled beta-agonists, leukotriene antagonists, leukotriene synthesis inhibitors, or any of their ingredients, including lactose and galactose
* clinically unstable disease of the ophthalmologic, neurological, hepatic, renal, connective tissue, genitourinary, gastrointestinal, cardiovascular or hematologic systems
* current cancer or history (within past ≤5 years) of cancer (except for successfully treated basal and squamous cell carcinomas of the skin); if cancer-free for >5 years, study participation may be allowed
* evidence of uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2012-08-23 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2014-07-08 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 576 randomized participants, 557 received treatment. The planned MK-1029 1 or 3 mg arm and the Montelukast + MK-1029 arm did not enroll any participants.
Groups:
- MK-1029 60 mg: Participants receive MK-1029 two 30 mg tablets QD for 12 weeks
- MK-1029 150 mg: Participants receive MK-1029 150 mg tablets QD for 12 weeks
- Montelukast 10 mg: Participants receive Montelukast 10 mg tablets QD for 12 weeks
- Placebo: Participants receive Placebo tablets QD for 12 weeks
- MK-1029 1 mg or 3 mg: Participants were to receive either MK-1029 1 mg or 3 mg tablets (dose to be determined based on results of interim analysis from Part I) QD. No participants were enrolled in this arm.
- Montelukast 10 mg + MK-1029: Participants were to receive Montelukast 10 mg tablets QD and MK-1029 tablets (dose to be determined based on results of interim analysis from Part I) QD. No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo | MK-1029 1 mg or 3 mg | Montelukast 10 mg + MK-1029
Started | 60 | 127 | 142 | 53 | 60 | 134 | 0 | 0
Treated Participants | 58 | 126 | 135 | 52 | 60 | 126 | 0 | 0
Completed | 43 | 93 | 106 | 41 | 46 | 94 | 0 | 0
Not Completed | 17 | 34 | 36 | 12 | 14 | 40 | 0 | 0
Not completed — Adverse Event | 1 | 14 | 5 | 4 | 5 | 7 | 0 | 0
Not completed — Lack of Efficacy | 1 | 8 | 6 | 1 | 1 | 6 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance with Study Drug | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 3 | 3 | 2 | 3 | 3 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 6 | 6 | 9 | 2 | 4 | 10 | 0 | 0
Not completed — Screen Failure | 2 | 1 | 7 | 1 | 0 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 2 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo | Total
Number analyzed (Participants) | 60 | 127 | 142 | 53 | 60 | 134 | 576
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (13.2) | 44.3 (12.4) | 43 (13.2) | 41.7 (12.2) | 43.7 (13.3) | 41.1 (12.4) | 42.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 78 | 77 | 31 | 32 | 47 | 298
  Male | 27 | 49 | 65 | 22 | 28 | 87 | 278
Asthma Phenotype [Number; unit: Participants] — The Asthma Phenotype in this study was defined as either "Th2-High" or "Th2-Low," based on measurements of asthmatic inflammation. Th2-High was defined according to the following 2 criteria at Visit 1: a peripheral-blood absolute eosinophil count ≥ 0.30 X 10^9/liters(L), and/or a peripheral-blood absolute eosinophil count ≥0.14 X 10^9/L with serum total IgE ≥100 IU/mL. Th2-Low was operationally defined as meeting neither of these criteria. Population: All participants who received ≥1 dose of study drug.
  Participants
    Th2-High: number analyzed (Participants) | 58 | 126 | 135 | 52 | 60 | 126 | 557
    Th2-High | 58 | 50 | 47 | 52 | 60 | 58 | 325
    Th2-Low | 0 | 76 | 88 | 0 | 0 | 68 | 232

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air (in liters) forcibly exhaled in one second. Repeated measurements of FEV1 were collected at visits during the 12 week active treatment period and the average change from baseline in FEV1 over the last 6 weeks of the 12-week-treatment period (visits at Week 6, Week 8, Week 10 and Week 12) was estimated using a constrained longitudinal data analysis (cLDA) model. In the cLDA analysis, baseline was the average FEV1 during the placebo run-in period and the post-baseline value was the average FEV1 over Week 6 to Week 12.
Time Frame: Baseline and last six weeks of treatment (visits at Week 6, Week 8, Week 10 and Week 12)
Population: T helper cell type 2 (TH2)-High participants who received ≥1 study drug dose and had FEV1 data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 57 | 50 | 47 | 52 | 60 | 58
Liters | 0.065 [-0.009 to 0.139] | 0.004 [-0.075 to 0.083] | 0.063 [-0.019 to 0.144] | 0.036 [-0.04 to 0.112] | 0.039 [-0.033 to 0.111] | 0.043 [-0.032 to 0.119]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in least squares (LS) means for average change from Baseline over Week 6 to Week 12 in FEV1: MK-1029 10 mg vs. Placebo. Constrained longitudinal data analysis (cLDA) model includes terms for visit as categorical variable, prior inhaled corticosteroid (ICS) use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.685, cLDA model; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.084 to 0.127]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in FEV1: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.477, cLDA model; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.149 to 0.07]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in FEV1: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.733, cLDA model; Mean Difference (Final Values) = 0.019, 95% CI 2-sided [-0.092 to 0.13]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in FEV1: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.89, cLDA model; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.115 to 0.1]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in FEV1: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.935, cLDA model; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.109 to 0.1]

2. Primary Outcome: Percentage of Participants Who Experience Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the study drug, is also an AE.
Time Frame: Up to 14 weeks
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 58 | 126 | 135 | 52 | 60 | 126
Percentage of participants | 44.8 | 48.4 | 47.4 | 53.8 | 56.7 | 57.9

3. Primary Outcome: Percentage of Participants Who Discontinue Study Due to AEs
Description: as for outcome 2
Time Frame: Up to 14 weeks
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 58 | 126 | 135 | 52 | 60 | 126
Percentage of participants | 1.7 | 10.3 | 3.7 | 7.7 | 8.3 | 5.6

4. Secondary Outcome: Percentage of Asthma Exacerbation Days
Description: An asthma exacerbation day was defined as a day with ANY of the following: a decrease from Baseline in morning (AM) Peak Expiratory Flow (PEF) of more than 20%, an AM PEF of less than 180 liters (L)/min, an increase in Short Acting Beta2 Agonist (SABA) use of more than 70% (and a minimum increase of at least 2 puffs), an increase from Baseline in Daytime Asthma Symptom Score of more than 50%, an overnight asthma symptom of: Awake "all night", or an asthma attack. Information on asthma exacerbation days was recorded throughout the study in the participant's electronic diary (e-Diary), and an Analysis of Variance (ANOVA) was used to calculate the average percentage of days with asthma exacerbations over Week 6 to Week 12.
Time Frame: Week 6 to Week 12
Population: TH2-High participants who received ≥1 study drug dose and had asthma exacerbation data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Asthma Exacerbation Days
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 44 | 39 | 37 | 46 | 47 | 39
Percentage of Asthma Exacerbation Days | 17.704 [10.657 to 24.75] | 15.812 [8.334 to 23.29] | 15.435 [7.752 to 23.118] | 20.238 [13.353 to 27.124] | 19.657 [12.845 to 26.47] | 24.904 [17.424 to 32.384]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for percent of asthma exacerbation day over Week 6 through Week 12: MK- 1029 10 mg vs. Placebo. Analysis of variance (ANOVA) model includes the terms for treatment groups and prior ICS use (Yes/No). Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.169, ANOVA; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-17.48 to 3.08]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for percent of asthma exacerbation day over Week 6 through Week 12: MK- 1029 30 mg vs. Placebo. ANOVA model includes the terms for treatment groups and prior ICS use (Yes/No). Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.092, ANOVA; Mean Difference (Final Values) = -9.092, 95% CI 2-sided [-19.67 to 1.485]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for percent of asthma exacerbation day over Week 6 through Week 12: MK- 1029 60 mg vs. Placebo. ANOVA model includes the terms for treatment groups and prior ICS use (Yes/No). Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.083, ANOVA; Mean Difference (Final Values) = -9.469, 95% CI 2-sided [-20.19 to 1.25]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for percent of asthma exacerbation day over Week 6 through Week 12: MK- 1029 150 mg vs. Placebo. ANOVA model includes the terms for treatment groups and prior ICS use (Yes/No). Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.367, ANOVA; Mean Difference (Final Values) = -4.666, 95% CI 2-sided [-14.83 to 5.501]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for percent of asthma exacerbation day over Week 6 through Week 12: Montelukast vs. Placebo. ANOVA model includes the terms for treatment groups and prior ICS use (Yes/No). Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.308, ANOVA; Mean Difference (Final Values) = -5.247, 95% CI 2-sided [-15.36 to 4.871]

5. Secondary Outcome: Average Change From Baseline in Daytime Symptom Score (DSS)
Description: The Daytime Symptom Score assessed daytime asthma symptoms. In the evening just before going to bed, participants scored their asthma symptoms for the period since arising by answering the following 4 questions in eDiaries: 1) How often did you experience asthma symptoms today?, 2) How much did your asthma symptoms bother you?, 3) How much activity could you do today? and 4) How often did your asthma affect your activities today? The 4 questions were scored on a 7-point scale (0=best to 6=worst) and averaged for a single score. The average change from baseline in DSS over the last 6 weeks of the 12-week-treatment period (visits at Week 6, Week 8, Week 10 and Week 12) was estimated using a cLDA model. In the cLDA analysis, baseline was the average DSS score during the placebo run-in period and the post-baseline value was the average DSS Score over Week 6 to Week 12.
Time Frame: Baseline and last six weeks of treatment (visits at Week 6, Week 8, Week 10 and Week 12)
Population: TH2-High participants who received ≥1 study drug dose and had DSS data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 45 | 41 | 40 | 49 | 49 | 43
Score on a scale | -0.398 [-0.612 to -0.184] | -0.134 [-0.358 to 0.091] | -0.364 [-0.591 to -0.137] | -0.120 [-0.325 to 0.086] | -0.411 [-0.617 to -0.206] | -0.276 [-0.495 to -0.056]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for average change from Baseline to Week 12 in DSS: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.429, cLDA model; Mean Difference (Final Values) = -0.122, 95% CI 2-sided [-0.427 to 0.182]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for average change from Baseline to Week 12 in DSS: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.370, cLDA model; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [-0.169 to 0.454]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for average change from Baseline to Week 12 in DSS: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK- 1029 or Montelukast); Test type: Superiority; p = 0.579, cLDA model; Mean Difference (Final Values) = -0.089, 95% CI 2-sided [-0.402 to 0.225]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for average change from Baseline to Week 12 in DSS: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.305, cLDA model; Mean Difference (Final Values) = 0.156, 95% CI 2-sided [-0.142 to 0.454]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for average change from Baseline to Week 12 in DSS: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.372, cLDA model; Mean Difference (Final Values) = -0.136, 95% CI 2-sided [-0.434 to 0.163]

6. Secondary Outcome: Average Change From Baseline in Use of Short-Acting Beta-Agonists (SABAs)
Description: Twice daily (upon arising and before going to sleep), participants recorded the total number of puff (actuations) of SABA used for asthma symptoms in their eDiaries. The number of SABA puffs used in one day was calculated based on eDiary entries as the sum of daytime and nighttime number of puffs of SABA. The average change from baseline over the last 6 weeks of the 12-week-treatment period (visits at Week 6, Week 8, Week 10 and Week 12) in the daily number of SABA puffs was estimated using a cLDA model. In the cLDA analysis, Baseline was the average number of SABA puffs used in one day during the placebo run-in period and the post-baseline value was calculated as the average number of SABA puffs used in one day over Week 6 to Week 12.
Time Frame: Baseline and last six weeks of treatment (visits at Week 6, Week 8, Week 10 and Week 12)
Population: TH2-High participants who received ≥1 study drug dose and had SABA usage data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of SABA Puffs
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 46 | 41 | 40 | 49 | 49 | 43
Number of SABA Puffs | -1.373 [-1.847 to -0.899] | -0.920 [-1.420 to -0.421] | -0.955 [-1.461 to -0.450] | -0.571 [-1.031 to -0.111] | -1.234 [-1.694 to -0.774] | -0.845 [-1.334 to -0.356]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in SABA use: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use(Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.114, cLDA model; Mean Difference (Final Values) = -0.528, 95% CI 2-sided [-1.184 to 0.128]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in SABA use: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.827, cLDA model; Mean Difference (Final Values) = -0.075, 95% CI 2-sided [-0.75 to 0.6]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in SABA use: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.75, cLDA model; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.789 to 0.569]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in SABA use: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.403, cLDA model; Mean Difference (Final Values) = 0.275, 95% CI 2-sided [-0.371 to 0.921]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in SABA use: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.237, cLDA model; Mean Difference (Final Values) = -0.389, 95% CI 2-sided [-1.035 to 0.257]

7. Secondary Outcome: Average Change From Baseline in Number of Nocturnal Awakenings
Description: The number of nights per week (between consecutive visits) that a participant awakened with asthma was based on eDiary entries and was calculated by dividing the number of nights a participant awakened with asthma (positive responses of once, more than once, awake "all night") by the total number of nights (all responses) and then multiplying by 7 (standardized to a 7-day period). The average change from baseline in number of nocturnal awakenings over the last 6 weeks of the 12-week-treatment period (visits at Week 6, Week 8, Week 10 and Week 12) was estimated using a cLDA model. In the cLDA analysis, baseline was the average number of nocturnal awakenings during the placebo run-in period and the post-baseline value was calculated as the average number of nocturnal awakenings over Week 6 to Week 12.
Time Frame: Baseline and last six weeks of treatment (visits at Week 6, Week 8, Week 10 and Week 12)
Population: TH2-High participants who received ≥1 study drug dose and had nocturnal awakening data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of awakenings
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 46 | 41 | 40 | 49 | 49 | 43
Number of awakenings | -1.277 [-1.861 to -0.692] | -0.900 [-1.518 to -0.282] | -1.286 [-1.912 to -0.661] | -1.277 [-1.844 to -0.710] | -1.107 [-1.674 to -0.540] | -1.036 [-1.639 to -0.432]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in nocturnal awakenings: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.565, cLDA model; Mean Difference (Final Values) = -0.241, 95% CI 2-sided [-1.066 to 0.583]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in nocturnal awakenings: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.754, cLDA model; Mean Difference (Final Values) = 0.135, 95% CI 2-sided [-0.713 to 0.983]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in nocturnal awakenings: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.563, cLDA model; cLDA model = -0.251, 95% CI 2-sided [-1.104 to 0.603]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in nocturnal awakenings: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.559, cLDA model; Mean Difference (Final Values) = -0.241, 95% CI 2-sided [-1.053 to 0.571]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in nocturnal awakenings: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.863, cLDA model; Mean Difference (Final Values) = -0.071, 95% CI 2-sided [-0.883 to 0.741]

8. Secondary Outcome: Average Change From Baseline in Morning/Evening Peak Expiratory Flow (AM/PM PEF)
Description: PEF was defined as a person's maximum speed (rate) of expiration as measured with a peak flow meter in liters per minute. Participants performed triplicate PEF measurements twice daily using a PEF meter, in the AM upon rising and in the PM immediately before study drug administration at bedtime. All three values were recorded and the average of the best morning PEF and the best evening PEF for each day (AM/PM) was determined through the e-Diary. The average change from Baseline in AM/PM PEF over the last 6 weeks of a 12-week treatment period (visits at Week 6, Week 8, Week 10 and Week 12) was estimated using a cLDA model. In the cLDA analysis, baseline was the average AM/PM PEF value during the placebo run-in period and the post-baseline value was calculated as the average AM/PM PEF over Week 6 to Week 12.
Time Frame: Baseline and last six weeks of treatment (visits at Week 6, Week 8, Week 10 and Week 12)
Population: TH2-High participants who received ≥1 study drug dose and had AM/PM PEF data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minutes
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 46 | 41 | 40 | 49 | 49 | 43
Liters/minutes | -1.857 [-16.13 to 12.413] | 3.850 [-11.26 to 18.960] | 7.174 [-8.124 to 22.472] | 2.713 [-11.12 to 16.543] | -4.005 [-17.83 to 9.825] | -2.401 [-17.16 to 12.357]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in AM/PM PEF: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.958, cLDA model; Mean Difference (Final Values) = 0.544, 95% CI 2-sided [-19.92 to 21.007]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in AM/PM PEF: MK- 1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.559, cLDA model; Mean Difference (Final Values) = 6.251, 95% CI 2-sided [-14.81 to 27.307]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in AM/PM PEF: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.374, cLDA model; Median Difference (Final Values) = 9.575, 95% CI 2-sided [-11.62 to 30.766]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in AM/PM PEF: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.618, cLDA model; Mean Difference (Final Values) = 5.114, 95% CI 2-sided [-15.04 to 25.272]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for average change from Baseline over Week 6 to Week 12 in AM/PM PEF: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.876, cLDA model; Mean Difference (Final Values) = -1.604, 95% CI 2-sided [-21.76 to 18.554]

9. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire With Standardised Activities [AQLQ(S)] Overall and Domain Scores
Description: The AQLQ(S) is a 32-item questionnaire with questions on 4 domains (asthma symptoms, activity limitation, emotional function and environmental stimuli) over the previous 2 weeks. Responses were scored on a 7-point scale (1=worst to 7=best). Each domain score is defined as the average score of all answered questions in that domain. The AQLQ(S) Overall Score is defined as the average of all available item scores (1=worst to 7=best). The changes from baseline are presented for the overall scores and the individual domain scores. Baseline was the last measurement taken prior to the first double-blind study drug. The ending values were calculated as the average AQLQ(S) Overall Score and domain scores at Week 12 of a 12-week treatment period. Statistical analyses are provided for the AQLQ(S) Overall Scores only.
Time Frame: Baseline and Week 12
Population: TH2-High participants who received ≥1 study drug dose and had AQLQ(S) data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 53 | 47 | 42 | 47 | 53 | 54
Score on a scale
  Overall Score | 0.533 (1.007) | 0.256 (0.997) | 0.696 (1.040) | 0.999 (1.255) | 0.736 (1.028) | 0.458 (1.176)
  Activity Domain: number analyzed (Participants) | 53 | 47 | 42 | 45 | 52 | 53
  Activity Domain | 0.46 (1.05) | 0.27 (0.98) | 0.62 (1.08) | 0.96 (1.32) | 0.66 (1.03) | 0.44 (1.18)
  Symptoms Domain: number analyzed (Participants) | 53 | 47 | 42 | 45 | 52 | 53
  Symptoms Domain | 0.59 (1.20) | 0.34 (1.24) | 0.80 (1.12) | 1.02 (1.25) | 0.83 (1.11) | 0.47 (1.29)
  Emotional Function Domain: number analyzed (Participants) | 53 | 47 | 42 | 45 | 52 | 53
  Emotional Function Domain | 0.55 (1.35) | 0.06 (1.17) | 0.75 (1.26) | 1.12 (1.62) | 0.70 (1.20) | 0.45 (1.37)
  Environmental Stimuli Domain: number analyzed (Participants) | 53 | 47 | 42 | 45 | 52 | 53
  Environmental Stimuli Domain | 0.53 (1.19) | 0.21 (0.90) | 0.54 (1.20) | 0.89 (1.47) | 0.70 (1.18) | 0.49 (1.43)
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in AQLQ(S) Overall Score: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.682, cLDA model; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.288 to 0.440]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in AQLQ(S) Overall Score: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.807, cLDA model; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.422 to 0.329]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in AQLQ(S) Overall Score: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.403, cLDA model; Mean Difference (Final Values) = 0.165, 95% CI 2-sided [-0.222 to 0.552]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in AQLQ(S) Overall Score: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.051, cLDA model; Mean Difference (Final Values) = 0.375, 95% CI 2-sided [-0.001 to 0.751]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in AQLQ(S) Overall Score: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Positive differences are in favor of the first treatment group in the comparison (MK- 1029 or Montelukast); Test type: Superiority; p = 0.086, cLDA model; Mean Difference (Final Values) = 0.319, 95% CI 2-sided [-0.045 to 0.683]

10. Secondary Outcome: Percentage of Participants With a ≥0.5 Change From Baseline in AQLQ(S) Overall and Domain Scores
Description: The AQLQ(S) is a 32-item questionnaire with questions on 4 domains (asthma symptoms, activity limitation, emotional function and environmental stimuli) over the previous 2 weeks. Responses were scored on a 7-point scale (1=worst to 7=best). Each domain score is defined as the average score of all answered questions in that domain. The AQLQ(S) Overall Score is defined as the average of all available item scores (1=worst to 7=best). The percentage of participants who experienced a ≥0.5 increase in AQLQ(S) Overall and Domain Scores at Week 12 compared to baseline was calculated using the Miettinen and Nurminen (MN) method. Statistical analyses are provide for the AQLQ(S) Overall Score response rate only.
Time Frame: Baseline and Week 12
Population: TH2-High participants who received ≥1 study drug dose and had AQLQ(S) data at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 53 | 47 | 42 | 45 | 52 | 53
Percentage of participants
  Overall Score | 48.99 | 40.49 | 57.22 | 64.48 | 64.08 | 46.14
  Activity Domain | 47.19 | 40.46 | 50.00 | 60.07 | 52.36 | 42.61
  Symptoms Domain | 52.59 | 42.63 | 59.66 | 57.76 | 64.08 | 48.13
  Emotional Function Domain | 56.19 | 31.95 | 62.10 | 57.76 | 53.91 | 49.90
  Environmental Stimuli Domain | 41.79 | 42.60 | 59.66 | 59.97 | 53.16 | 48.13
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference for AQLQ(S) Response Rate: MK-1029 10 mg vs. Placebo. P-values, estimates and 95% confidence intervals (CIs) are based on the Miettinen and Nurminen (MN) method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.7687, MN method; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-16.0 to 21.3]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference for AQLQ(S) Response Rate: MK-1029 30 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.4943, MN Method; Mean Difference (Final Values) = -6.6, 95% CI 2-sided [-24.9 to 12.2]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference for AQLQ(S) Response Rate: MK-1029 60 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.3003, MN method; Mean Difference (Final Values) = 10.5, 95% CI 2-sided [-9.4 to 29.6]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference for AQLQ(S) Response Rate: MK-1029 150 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.0774, MN method; Mean Difference (Final Values) = 17.5, 95% CI 2-sided [-1.9 to 35.7]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference for AQLQ(S) Response Rate: Montelukast vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.0555, MN method; Mean Difference (Final Values) = 18.2, 95% CI 2-sided [-0.4 to 35.5]

11. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Score
Description: The ACQ is a validated 6-item measure of asthma control to evaluate asthma control in response to therapy. Participants evaluate their asthma over the previous week by answering 6 questions: How often were you woken by your asthma during the night? How bad were your asthma symptoms when you woke up in the morning? How limited were you in your activities because of your asthma? How much shortness of breath did you experience because of your asthma? How much of the time did you wheeze? How many puffs/inhalations of short-acting bronchodilator have you used each day? Each response to a question was scored on a 7-point scale (0=best to 6=worst). The ACQ score is the average of the scores for the 6 items. Change from baseline to Week 12 in ACQ was estimated using a cLDA model. In the cLDA analysis, the Baseline value was the last measurement taken prior to the first double-blind study drug and the post-baseline value was calculated as the average ACQ Score at Week 12.
Time Frame: Baseline and Week 12
Population: TH2-High participants who received ≥1 study drug dose and had ACQ data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 53 | 47 | 42 | 47 | 52 | 54
Score on a scale | -0.807 [-1.088 to -0.527] | -0.736 [-1.033 to -0.438] | -0.855 [-1.170 to -0.541] | -1.066 [-1.364 to -0.768] | -0.931 [-1.215 to -0.648] | -0.704 [-0.982 to -0.426]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in ACQ Score: MK-1029 10 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.603, cLDA model; Mean Difference (Final Values) = -0.104, 95% CI 2-sided [-0.495 to 0.288]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in ACQ Score: MK-1029 30 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.875, cLDA model; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.436 to 0.372]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in ACQ Score: MK-1029 60 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.476, cLDA model; Mean Difference (Final Values) = -0.151, 95% CI 2-sided [-0.568 to 0.265]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in ACQ Score: MK-1029 150 mg vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.079, cLDA model; Mean Difference (Final Values) = -0.362, 95% CI 2-sided [-0.767 to 0.042]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for change from Baseline to Week 12 in ACQ Score: Montelukast vs. Placebo. cLDA model includes terms for visit as categorical variable, prior ICS use (Yes/No) and treatment by visit. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.257, cLDA model; Mean Difference (Final Values) = -0.227, 95% CI 2-sided [-0.621 to 0.166]

12. Secondary Outcome: Percentage of Participants With a ≥0.5 Change From Baseline in ACQ Score
Description: The ACQ is a validated 6-item measure of asthma control to evaluate asthma control in response to therapy. Participants evaluate their asthma over the previous week by answering 6 questions: How often were you woken by your asthma during the night? How bad were your asthma symptoms when you woke up in the morning? How limited were you in your activities because of your asthma? How much shortness of breath did you experience because of your asthma? How much of the time did you wheeze? How many puffs/inhalations of short-acting bronchodilator have you used each day? Each response to a question was scored on a 7-point scale (0=best to 6=worst). The ACQ score is the average of the scores for the 6 items. The percentage of participants who experienced a ≥0.5 decrease in ACQ Score at Week 12 compared to Baseline was calculated using the MN method.
Time Frame: Baseline and Week 12
Population: TH2-High participants who received ≥1 study drug dose and had ACQ data at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 53 | 47 | 42 | 45 | 51 | 54
Percentage of participants | 65.51 | 59.57 | 66.60 | 71.11 | 64.72 | 62.43
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference for change from Baseline to Week 12 in ACQ response rate: MK-1029 10 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.742, MN method; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-15.1 to 21.1]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference for change from Baseline to Week 12 in ACQ response rate: MK-1029 30 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.7248, MN method; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-22.1 to 15.4]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference for change from Baseline to Week 12 in ACQ response rate: MK-1029 60 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.6991, MN method; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-15.6 to 22.6]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference for change from Baseline to Week 12 in ACQ response rate: MK-1029 150 mg vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.3934, MN method; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [-10.6 to 26.2]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference for change from Baseline to Week 12 in ACQ response rate: Montelukast vs. Placebo. P-values, estimates and 95% CIs are based on the MN method stratified by prior ICS use (Yes/No); Test type: Superiority; p = 0.8032, MN method; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-16.0 to 20.5]

13. Secondary Outcome: Percentage of Asthma Attack Days
Description: An asthma attack was defined as asthma symptoms during the previous 24 hours requiring one or more of the following: corticosteroid use (systemic), unscheduled visit to the doctor or urgent care clinic, unscheduled visit to the emergency department or hospitalization. Information on asthma attacks was recorded throughout the study in the participant's e-Diary, and an Analysis of Variance (ANOVA) was used to calculate the average percentage of asthma attack days over Week 6 to Week 12 of a 12-week treatment period.
Time Frame: Week 6 to Week 12
Population: TH2-High participants who received ≥1 study drug dose and had asthma attack data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 43 | 39 | 37 | 45 | 47 | 39
Percentage | 0.482 [-0.159 to 1.122] | 0.182 [-0.49 to 0.854] | 0.017 [-0.673 to 0.708] | 0.637 [0.011 to 1.262] | 0.248 [-0.364 to 0.86] | 0.557 [-0.115 to 1.230]
Statistical Analysis 1: Comparison: MK-1029 10 mg vs Placebo; Difference in LS means for percent of asthma attack days over Week 6 to Week 12 of a 12-week treatment period: MK-1209 10 mg vs. Placebo. ANOVA model includes terms for prior ICS use (Yes/No) and treatment. Negative differences are in favor of the first treatment group in the comparison (MK- 1029 or Montelukast); Test type: Superiority; p = 0.873, ANOVA; Mean Difference (Final Values) = -0.075, 95% CI 2-sided [-1.004 to 0.853]
Statistical Analysis 2: Comparison: MK-1029 30 mg vs Placebo; Difference in LS means for percent of asthma attack days over Week 6 to Week 12 of a 12-week treatment period: MK-1209 30 mg vs. Placebo. ANOVA model includes terms for prior ICS use (Yes/No) and treatment. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.437, ANOVA; Mean Difference (Final Values) = -0.376, 95% CI 2-sided [-1.326 to 0.575]
Statistical Analysis 3: Comparison: MK-1029 60 mg vs Placebo; Difference in LS means for percent of asthma attack days over Week 6 to Week 12 of a 12-week treatment period: MK-1209 60 mg vs. Placebo. ANOVA model includes terms for prior ICS use (Yes/No) and treatment. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.270, ANOVA; Mean Difference (Final Values) = -0.540, 95% CI 2-sided [-1.504 to 0.423]
Statistical Analysis 4: Comparison: MK-1029 150 mg vs Placebo; Difference in LS means for percent of asthma attack days over Week 6 to Week 12 of a 12-week treatment period: MK-1209 150 mg vs. Placebo. ANOVA model includes terms for prior ICS use (Yes/No) and treatment. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.865, ANOVA; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.839 to 0.997]
Statistical Analysis 5: Comparison: Montelukast 10 mg vs Placebo; Difference in LS means for percent of asthma attack days over Week 6 to Week 12 of a 12-week treatment period: Montelukast vs. Placebo. ANOVA model includes terms for prior ICS use (Yes/No) and treatment. Negative differences are in favor of the first treatment group in the comparison (MK-1029 or Montelukast); Test type: Superiority; p = 0.503, ANOVA; Mean Difference (Final Values) = -0.309, 95% CI 2-sided [-1.219 to 0.600]

ADVERSE EVENTS:
Time Frame: Up to 14 weeks (Up to 2 weeks after last dose of study drug)
Description: The safety population consisted of all randomized participants who received ≥1 dose of study drug.
Arm/Group | MK-1029 10 mg | MK-1029 30 mg | MK-1029 60 mg | MK-1029 150 mg | Montelukast 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/126 | 0/135 | 0/52 | 0/60 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/58 | 2/126 | 2/135 | 1/52 | 0/60 | 1/126
Other Adverse Events (participants affected / at risk) | 15/58 | 24/126 | 27/135 | 19/52 | 19/60 | 42/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1029 10 mg (N=58) | MK-1029 30 mg (N=126) | MK-1029 60 mg (N=135) | MK-1029 150 mg (N=52) | Montelukast 10 mg (N=60) | Placebo (N=126)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kaposi's varicelliform eruption (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1029 10 mg (N=58) | MK-1029 30 mg (N=126) | MK-1029 60 mg (N=135) | MK-1029 150 mg (N=52) | Montelukast 10 mg (N=60) | Placebo (N=126)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 10 (10) | 7 (7) | 5 (5) | 12 (12)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 7 (10) | 1 (1) | 2 (3) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 15 (19) | 5 (5) | 8 (8) | 11 (12) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.